CLINICAL TRIAL: NCT01864616
Title: The Impact of Vitamin D on Disease Activity in Crohn's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We couldn't recruit the sample the we required
Sponsor: University of Saskatchewan (Other)
Collaborators: Dania Alrefai (Unknown); Dr.Jennifer Jones (Unknown); Dr.Hani Jawa (Unknown); Dr.Wael El-matary (Unknown); Saudi Arabian Cultural Bureau (Unknown)
Responsible Party: Principal Investigator, Hassanali Vatanparast, Associate Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VCD-060
Record Dates: First submitted 2013-05-22; First posted 2013-05-29 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Crohn Disease
Keywords: Vitamin D; Crohn disease; Disease activity; Inflammation; prevention
MeSH Terms: conditions — Crohn Disease; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 3 (Experimental): Vitamin D3, 10,000 IU daily
  Interventions: Dietary Supplement: Vitamin D3
- Group 2 (Experimental): Vitamin D3 2,000 IU daily
  Interventions: Dietary Supplement: Vitamin D3
- Group 1 (Experimental): Vitamin D3 600 IU daily (Control group, RDA level)
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3

SUMMARY:
The purpose for this study is to determine the effect of vitamin D supplementation on disease activity in Crohn's disease patients in Canada and Saudi Arabia

DETAILED DESCRIPTION:
Hypothesis 1: Patients who are suffering from Crohn's disease are at risk of vitamin D deficiency.

To determine vitamin D status and disease activity in Crohn's disease cases in Canada and Saudi Arabia.

Hypothesis 2: Providing vitamin D in doses higher than RDA (Recommended Dietary Allowance) reduces disease activity in Crohn's disease cases.

To evaluate the impact vitamin D in doses higher than RDA (Recommended Dietary Allowance) on disease activity in Crohn's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosis with an active Crohn's disease,
* age above of 16 years

Exclusion Criteria:

* remission or the duration of disease is more than 2 years,
* pregnancy,
* liver or kidney failure,
* inability to take oral supplements or medicine

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The changes in disease activity on groups | (0), 5 weeks, 9 weeks, after 2 months
  We have 4 time points, baseline (0), Week 5, Week 9 (termination) and Week 17 (follow up) To measure the disease activity, we will examine C- reactive protein levels "blood test", Fecal fat " stool test" and Crohn's disease activity index (CDAI)"tool".

SECONDARY OUTCOMES:
nutritional status | 0, 5 weeks, 9 weeks, 2 months later
  We have 4 time points, baseline (0), Week 5, Week 9 (termination) and Week 17 (follow up). We will use 24-hour dietary recalls for 9 different days.
vitamin D status | (0), Week 5, Week 9 (termination) and 2 months later
  We have 4 time points, baseline (0), Week 5, Week 9 (termination) and Week 17 (follow up) vitamin D status: Blood test
Health related quality of life | (0), Week 5, Week 9 (termination) and 2 months later (follow up)
  We have 4 time points, baseline (0), Week 5, Week 9 (termination) and Week 17 (follow up). We will use Health related quality of life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hassanali Vatanparast, MD,PhD, Principal Investigator — University of Saskatchewan, Saskatoon, SK,Canada; Jennifer Jones, MD,MSc,FRCPC, Study Director — Royal University Hospital, Saskatoon, Saskatchewan, Canada; Hani Jawa, MBBS,ABIM,FRCPC, Study Director — King Abdulaziz University, jeddah, Saudi Arabia; Wael El-matary, MBChB,MSc,MD,FRCPCH, Study Director — University of Manitoba; Dania Alrefai, M.Sc, Principal Investigator — University of Saskatchewan
Locations (2):
- IBD clinic; Royal University Hospital, Saskatoon, Saskatchewan, Canada
- Internal Medicine Department; King Abdulaziz University Hospital, Jeddah, Saudi Arabia